CLINICAL TRIAL: NCT02736877
Title: Corneal Transplantation Guided by OCT RESCAN: Pre-op, Intra-op and Post-op Evaluation
Brief Title: Corneal Transplantation Guided by OCT RESCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Eye Clinic Day Hospital, São Paulo (Other)
Responsible Party: Principal Investigator, Walton Nose, Professor of Ophthalmology, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCAN2016
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Cornea; Keratoconus; Bullous Keratopathy; Corneal Dystrophy
Keywords: keratoconus; bullous keratopathy; corneal dystrophy
MeSH Terms: conditions — Corneal Diseases; Keratoconus; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumera Microscope with OCT RESCAN (Experimental): In the group microscope coupled to OCT, patients will undergo corneal surgery using the Lumera Microscope WITH RESCAN OCT - ZEISS. The team of surgeons will answer the questionnaire on the surgical difficulty regarding corneal transplantation
  Interventions: Procedure: Lumera Microscope with OCT RESCAN
- Conventional Microscope (Active Comparator): The control group will undergo corneal transplant with conventional microscope without coupled OCT. The team of surgeons will answer the questionnaire on the surgical difficulty regarding corneal transplantation
  Interventions: Procedure: Conventional Microscope

INTERVENTIONS:
Procedure: Lumera Microscope with OCT RESCAN — corneal transplantation guided by Lumera Microscope with OCT RESCAN
  Arms: Lumera Microscope with OCT RESCAN
Procedure: Conventional Microscope — corneal transplantation guided by Conventional Microscope
  Arms: Conventional Microscope

SUMMARY:
The investigators will evaluate 30 patients with surgical indication for corneal transplantation. Participants will be divided according to the following diseases diseases: keratoconus, bullous keratopathy, corneal dystrophies. Participants will be informed about the risks and benefits of the study and sign an informed consent form. In the preoperative evaluation will be submitted to a complete ophthalmologic examination with complementary tests, such as optical coherence tomography.

One group of participants will undergo corneal surgery using the OCT Lumera microscope RESCAN - ZEISS and another group with a conventional microscope. Everyone will have their filmed and documented surgery. The team of surgeons will answer the questionnaire on the surgical difficulty about the ease of assessing corneal transplantation. After surgery, participants will be assessed on days 1, 7,15, 30, 60, 90 and 180 after surgery.

Surgeries and study procedures will be performed by the same team of surgeons and performed by IPEPO - Paulista Institute of Studies and Research in Ophthalmology / Vision Institute.

DETAILED DESCRIPTION:
Participants will be allocated in one of the following groups:

1. Control Group The control group will undergo corneal transplant with conventional microscope without coupled OCT. The team of surgeons will answer the questionnaire on the surgical difficulty regarding corneal transplantation (ANNEX 1).
2. Group OCT RESCAN In the group microscope coupled to OCT, patients will undergo retinal surgery using the Lumera Microscope WITH RESCAN OCT - ZEISS. The team of surgeons will answer the questionnaire on the surgical difficulty regarding corneal transplantation (ANNEX 1).

The investigators will evaluate intraoperative conditions, complications, operative time and postoperative results in both groups.

All patients will be monitored and evaluated with full ophthalmological examination in all postoperative visits (day 1, 7,15,30, 60, 90, 180) and will be subjected to the following tests:

* Measurement of visual acuity with best correction
* Previous Biomicroscopy
* Corneal Topography
* tonometry
* Optical coherence tomography (OCT)
* Microscopy speculate

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity less than 20/60 in the affected eye
* 18 years at least
* Diagnostic of the following diseases:

  * keratoconus
  * Keratopathy Bullosa
  * Corneal dystrophy

Exclusion Criteria:

* Better visual acuity than or equal to 20/60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Assess optimal maneuvers in corneal transplantation (separation layers) | Day 0
  assessed by a questionnaire responded by surgeons (no difficulty, some difficulty, very difficulty)

SECONDARY OUTCOMES:
Compare the time of surgery between groups | Day 0
  by a questionnaire responded by surgeons (until 30 minutes, between 30-60 minutes, more than 60 minutes)
To describe the surgical difficulty for corneal transplantation | Day 0
  by a questionnaire responded by surgeons (no difficulty, some difficulty, very difficulty)
Change of Day 1 Ocular inflammation at 1 month (Day 30) | from Day1 to Day30
  ocular inflammation scored as mild, moderate or severe
Change from Baseline Intraocular Pressure at 6 months (Day180) | from Baseline to Day 180
  intraocular pressure assessed by goldmann tonometer
Change from Baseline Visual Acuity at 6 months (Day 180) | from Baseline to Day 180
  visual acuity tested by ETDRS chart

CONTACTS AND LOCATIONS:
Overall Officials: Walton Nose, MD, PhD, Principal Investigator — Federal University of São Paulo UNIFESP

IPD SHARING:
Plan to Share IPD: Yes
scientific publication